CLINICAL TRIAL: NCT00548483
Title: Phase 2 Study of Comparison of High Dose and Low Dose Dexamethasone in Preventing Post-Extubation Airway Obstruction in Adults
Brief Title: Comparison of High Dose and Low Dose Dexamethasone in Preventing Post-Extubation Airway Obstruction in Adults
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Chao-Hsien, Lee, Mackay memorial hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MMH-I-S-107
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Airway Obstruction
Keywords: Endotracheal intubation; Laryngeal edema; Cuff-leak test; Corticosteroids; This study was to ascertain whether administration of dexamethasone to critically intubated patients prevent postextubation airway obstruction.; This study was to compare high dose and low dose dexamethasone in preventing noninvasive ventilation or reintubation among critically ill intubated patients
MeSH Terms: conditions — Airway Obstruction; Laryngeal Edema | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): dexamethasone 5mg was administered every 6 hour for 1 day
  Interventions: Drug: dexamethasone (Oradexon, Nederland)
- 2 (Active Comparator): dexamethasone 10mg was administered every 6 hour for 1 day
  Interventions: Drug: dexamethasone (Oradexon, Nederland)

INTERVENTIONS:
Drug: dexamethasone (Oradexon, Nederland) — dexamethasone 5mg was administered every 6 hour for 1 day in group 1 and dexamethasone 10mg was administered every 6 hour for 1 day in group 2

SUMMARY:
The specific objectives were to determine whether high dose dexamethasone are more effective than low dose dexamethasone in the reduction or prevention of post-extubation airway obstruction among patients with a cuff leak volume (CLV) < 110 mL.

DETAILED DESCRIPTION:
Controversy currently exists regarding the effectiveness of prophylactic steroid therapy for patients considered at high risk for post-extubation stridor. Studies regarding the efficacy of prophylactic corticosteroids for intubated patients have yielded conflicting results due to differences in the number, dose, or type of corticosteroids administered.

Only a limited number of prospective trials involving adults and evaluating the benefits and the dose of corticosteroid therapy prior to extubation have been conducted.The present study was conducted to evaluate the effects of prophylactic dexamethasone therapy for a subset of high-risk patients who had been intubated for > 48 hours and who were undergoing their first elective extubation in an ICU setting.

ELIGIBILITY:
Inclusion Criteria:

All patients were > 18 years of age and met the following weaning criteria:

1. Temperature ≤ 38°C for > 8 hours,
2. Discontinuous use of sedatives,
3. Heart rate ≥ 70 and ≤ 130 /min,
4. Systolic blood pressure (SBP) ≥ 80 mm Hg in the absence of vasopressors,
5. Fraction of inspired oxygen (FiO2) ≤ 0.6, PaO2 ≥ 60, and partial pressure of oxygen (PaO2)/FiO2 ratio > 200,
6. Positive end-expiratory pressure (PEEP) ≤ 5 cm H2O,
7. Rapid and shallow ratio of frequency to tidal volume (f/VT ≤ 105),
8. Minute ventilation ≤ 15 L/min, and
9. pH ≥ 7.3. Supplemental oxygen was continued to maintain an oxygen saturation > 95% as measured by a pulse oximeter.

Exclusion Criteria:

1. A history of extubation during the same hospitalization
2. Administration of corticosteroids seven days prior to extubation.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-04; Primary Completion 2008-03 (Estimated); Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
absolute cuff leak volumes and relative cuff leak volume to tidal volume(%)(measured CLV-baseline CLV) X 100/ tidal volume) | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Hsien Lee, MD, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- No. 92, SEC. 2, CHUNG SHAN N. RD, TAIPEI, TAIWAN., Taipei, Taiwan

REFERENCES:
- [Background] Lee CH, Peng MJ, Wu CL. Dexamethasone to prevent postextubation airway obstruction in adults: a prospective, randomized, double-blind, placebo-controlled study. Crit Care. 2007;11(4):R72. doi: 10.1186/cc5957. PMID 17605780
- [Background] Cheng KC, Hou CC, Huang HC, Lin SC, Zhang H. Intravenous injection of methylprednisolone reduces the incidence of postextubation stridor in intensive care unit patients. Crit Care Med. 2006 May;34(5):1345-50. doi: 10.1097/01.CCM.0000214678.92134.BD. PMID 16540947
- [Background] Francois B, Bellissant E, Gissot V, Desachy A, Normand S, Boulain T, Brenet O, Preux PM, Vignon P; Association des Reanimateurs du Centre-Ouest (ARCO). 12-h pretreatment with methylprednisolone versus placebo for prevention of postextubation laryngeal oedema: a randomised double-blind trial. Lancet. 2007 Mar 31;369(9567):1083-9. doi: 10.1016/S0140-6736(07)60526-1. PMID 17398307